CLINICAL TRIAL: NCT01919645
Title: Effectiveness and Safety of Physical Exercises in the Improvement of the Sleep Quality in Women With Rheumatoid Arthritis: A Randomized Clinical Trial Study
Brief Title: Effectiveness and Safety of Physical Exercises in the Improvement of the Sleep Quality. Regarding Rheumatoid Arthritis
Acronym: SRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Andrea Kayo, PhD Student, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHK2013
Record Dates: First submitted 2013-08-03; First posted 2013-08-09 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Sleep Disorders; Polysomnography; Sleep Stages; Physical Exercise
MeSH Terms: conditions — Arthritis, Rheumatoid; Sleep Wake Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined Training Group (Experimental): Combined Training - (strength + aerobics).
  A combined training (CT)is performed, having aerobics exercises (AE)using a stationary bicycle and strength training in workout devices.
  The strength training (ST) will be performed by isotonic exercises recruiting the main muscle groups. They exercises are: Chest Press, Leg Press, Vertical Traction, Leg Extension and Abdominal Crunch.
  Interventions: Other: Combined Training ( Strength + Aerobics)
- Control Group (Placebo Comparator): The control group patients did not perform any intervention through physical exercises. They were oriented on Sleep Hygiene and were followed during the study. They were asked to come to the following visits (at weeks 8 and 16) and to 2 additional visits to get and then return the actigraph. During this period, they were followed through phone calls once a month and were asked for sleep hygiene and were reminded of their assessment dates.
  Interventions: Other: Combined Training ( Strength + Aerobics)

INTERVENTIONS:
Other: Combined Training ( Strength + Aerobics) — Strength training performed using workout devices and aerobic training performed using stationary bicycle.

SUMMARY:
Physical exercise programs are effective and safe for the improvement of the sleep efficiency in patients with Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

• Women ages 35-65 years diagnosed with Rheumatoid Arthritis according with the American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR)Criteria; Pittsburgh Sleep Quality Index ≥ 5; electrocardiogram test (ECG) at rest and at regular effort.

Exclusion Criteria:

* Patients with joint restrictions due to disease.
* Other rheumatoid-associated diseases (Fibromyalgia) with the exception of Osteoarthritis of low degree.
* Those who are uncontrollably hypertense, diabetic, with thyroidopathy and cardiorespiratory diseases which stop them from practicing exercises.
* Class II obesity (IMC ≥ 35 Kg/m2).
* Cognitive deficits.
* Depression.
* Patients not following the study rules such as exercise hours and / or time for the proposed program.
* Current physical exercise practitioner.
* Those undergoing medication treatment which would interfere sleep.
* Night shift workers who disrespect regular working schedule.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Improvement of sleep through a polysomnogram exam. | at baseline and at end-week 16
  Evaluation of N3 stage of the sleep through a polysomnogram before and after 16 weeks of supervised exercises.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea H Kayo, PHD student, Principal Investigator — Federal University of São Paulo
Locations (1):
- Centro de Estudos em Psicobiologia e Exercício (CEPE) da Associação Fundo de Incentivo a Pesquisa (AFIP), São Paulo, São Paulo, Brazil